CLINICAL TRIAL: NCT03777124
Title: Phase II Study of SHR-1210(Anti-PD-1 Antibody) Combination With Apatinib Versus Pemetrexed and Carboplatin in Subjects With KRAS Mutant Stage IV Non-squamous Non-small Cell Lung Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The sponsor's R&D strategy is adjusted.
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Collaborators: Shanghai Chest Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHR-1210-II-214
Record Dates: First submitted 2018-12-13; First posted 2018-12-17 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: NSCLC Stage IV; KRAS Gene Mutation; PD-1 Antibody; Chemotherapy Effect
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — camrelizumab; apatinib; Pemetrexed; Carboplatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SHR-1210 +apatinib (Experimental): subject will receive SHR-1210 200mg every 2 weeks, apatinib 250mg every day
  Interventions: Drug: SHR-1210; Drug: Apatinib
- chemotherapy (Active Comparator): Pemetrexed 500mg/m2, Day 1 of each 21 day, 4 cycles carboplatin AUC 5 on Day 1 of each 21 day, 4 cycles followed by pemetrexed 500mg/m2 until progression Q3W
  Interventions: Drug: Pemetrexed; Drug: Carboplatin

INTERVENTIONS:
Drug: SHR-1210 — Subjects receive SHR-1210 intravenous every 2 weeks
  Arms: SHR-1210 +apatinib
Drug: Apatinib — Subjects receive Apatinib orally every day
  Arms: SHR-1210 +apatinib
Drug: Pemetrexed — Subjects receive Pemetrexed intravenous every 3 weeks
  Arms: chemotherapy
Drug: Carboplatin — subjects receive carboplatin intravenous every 3 weeks
  Arms: chemotherapy

SUMMARY:
This is a randomized, open-label, multi-center, phase II trial to evaluate the efficacy and safety of SHR-1210 plus apatinib mesylate versus Pemetrexed and Carboplatin in Subjects with KRAS mutant stage IV non-squamous Non-small Cell Lung Cancer

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with histopathological diagnosis of adenocarcinoma non-small cell lung cancer (NSCLC) and clinical stage IV
2. has not received prior systemic treatment for metastatic NSCLC.
3. Has a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) Performance Status
4. confirmes by the central laboratory as KRAS gene mutation
5. Has archived Tumor tissue samples
6. Subject must have a measurable target lesion based on RECIST v1.1 .
7. Women of childbearing age must undergo a serological pregnancy test within 3 days before the first dose with negative results. Female subjects of reproductive age and male subjects whose spouse is a woman of reproductive age must agree to effective contraception within 180 days after the study period and the last dose of the study drug.
8. Subjects should be voluntarily participate in clinical studies and informed consent should be signed.

Exclusion Criteria:

1. active brain metastases and meningeal metastasis
2. uncontrollable tumor-related pain
3. massive pleural effusion, peritoneal effusion or pericardial effusion which cannot be controlled by repeated drainage;
4. radiotherapy to lung that is >30 Gy within 24 weeks before the first dose,
5. imaging (CT or MRI) showed that the tumor invading the large vessels
6. Known EGFR/ALK mutation.
7. subjects with any known or suspected autoimmune diseases
8. subjects with known or suspected interstitial pneumonia;
9. Subjects with severe cardiovascular and cerebrovascular diseases
10. arteriovenous thrombosis events, such as deep vein thrombosis and pulmonary embolism, occurred within 3 months;
11. female subjects who are pregnant or lactation or who plan to be pregnant during the study period;
12. positive HIV test;
13. active hepatitis B
14. evidence of active TB infection within 1 year before first dose;
15. severe infection occurred within 4 weeks before the first dose
16. patients with clinically significant bleeding symptoms or with obvious bleeding tendency in the first month
17. subjects who is on systemic immunogenic agents;
18. a history of severe allergic reactions to other monoclonal antibodies/fusion proteins;
19. History of severe allergic reactions to carboplatin or pemetrexed or their preventive drugs;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — KRAS mutant
Enrollment: 25 (Actual)
Dates: Start 2019-07-11 (Actual); Primary Completion 2023-06-29 (Actual); Study Completion 2023-06-29 (Actual)

PRIMARY OUTCOMES:
Duration of Progression-Free Survival (PFS) as Assessed by the Independent Review Committee Using RECIST v1.1 | up to approximately 40 months
  PFS, defined as the time from randomization to the first occurrence of disease progression as determined by the Independent Review Committee Using RECIST v1.1 or death from any cause, whichever occurs first. Patients who have not experienced disease progression or death at the time of analysis will be censored at the time of last tumor assessment.

SECONDARY OUTCOMES:
Duration of Progression-Free Survival (PFS) as Assessed by the Investigator Using RECIST v1.1 | up to approximately 40 months
  Time Frame: Baseline until PD or death, whichever occurs first
Duration of Overall Survival (OS) | up to approximately 40 months
  Baseline until death from any cause
Objective Response Rate (ORR) | up to approximately 40 months
  The percentage of patients with CR and PR assessed by investigators according to Recist v 1.1.
disease control rate (DCR) | up to approximately 40 months
  The proportion of patients who have achieved complete response， partial response and Stable disease assessed by investigators according to Recist v 1.1.
Duration of response （DoR） | up to approximately 40 months
  Duration of response （DoR）
Adverse events (AEs) | up to approximately 40 months
  All adverse event/Serious adverse event that occurred during the study period according to CTCAE v 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Jianjun Zou, MD, PhD, Study Director — Jiangsu HengRui Medicine Co., Ltd.; Shun Lu, MD, PhD, Principal Investigator — Jiaotong University,Shanghai chest Hospital
Locations (1):
- Shanghai Chest Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided